CLINICAL TRIAL: NCT01671293
Title: Remote Care Model for Supporting Prediabetes Patients
Brief Title: Multicomponent Telecare Model for Supporting Prediabetes Patients
Acronym: MTELECAREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: National Fund for Research and Development in Health, Chile (Other); Corporación Municipal de Educación, Salud y Recreación de La Florida (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FONIS SA10I20017
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Prediabetic State; Glucose Intolerance
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multicomponent remote care model (Experimental): A remote intervention based on counseling (telephone-based).
  Interventions: Behavioral: Multicomponent remote care model
- Usual care (Active Comparator): Usual care.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Multicomponent remote care model — A remote intervention based on counseling (telephone-based) was implemented. This counseling intervention is the core of the multi-component model, which also includes counseling through text messages, the purveyance of educational material, and self-monitoring equipment (pedometer & waist circumference measuring tape). The phone counseling is made by health centers professionals who have been trained to apply theories on behavioral change and decision-making. Phone counseling is conducted at least once a month. Messages are sent weekly and are related to the topics referred to in phone counseling sessions. The educational material and equipment -respectively- seek to provide additional information and foster the habit of self-monitoring progress and/or reversions in the change process.
  Arms: Multicomponent remote care model
Other: Usual care — Usual care from health centers consisting of medical indication of physical activity and healthy eating recommendations, as well as referral to Dietitian if appropriate, an invitation to participate in educational activities at health centers and periodic inspection appointments
  Arms: Usual care

SUMMARY:
The purpose of this study is to determine whether a multi-component remote care model (telephone-based) is effective to achieve the modification of unhealthy eating practices and increase physical activity in adults who have prediabetes and over-weight/obesity. The effectiveness of the remote care model will be determined with respect to the mentioned practices as well as anthropometric parameters (Waist circumference and Weight) and clinical parameters (Fasting Glucose, Triglycerides, Total Cholesterol) which are sensitive to changes in these habits. The counseling intervention is the core of the multi-component tele-care model, which also includes counseling-through text messages, supply of Educational material and self-monitoring equipment (pedometers and measuring tape for patients to check their waist circumference).

DETAILED DESCRIPTION:
International data report that the population with prediabetes is approximately twice the population with Diabetes Mellitus type 2 (DM2) both in the U.S. and Latin America. Given prediabetes estimated prevalence in Chile (8 to 15%) and considering the high risk for developing DM2 that prediabetic people present, as well as the high cost associated with treating this disease and its consequences, it is essential to look for strategies to prevent and/or delay this process. People under 45 years who are overweight and have altered glucose tolerance test constitute a population who is at high risk for developing DM2 (MINSAL, 2009). It has been shown that weight loss and increase of moderate physical activity reduces by 58% the risk of developing DM2 (The Diabetes Prevention Program Research Group, 2002), however, at primary care, people who are informed of having prediabetes usually present no access to the available services to support them in the process of changing behaviors that are at the core of this condition.

This study aims to design, implement and evaluate a multi-component remote care model to support people with prediabetes who are overweight or obese, at self-management of their risk behaviors of unhealthy diet and physical inactivity. This study seeks to determine whether remote care interventions aimed at overweight or obese people with prediabetes, carried out by professionals trained in motivational interviewing, behavior change theories and support health decision-making, with knowledge of prediabetes and effective interventions for coping are effective for: a) Increase participants knowledge about the risks of this condition and how to prevent them b) Provide effective support that results in an increase in daily physical activity c) Provide effective support to ensure change in their eating habits d) Achieve reduction in clinical parameters values of glucose, cholesterol and triglycerides e) Attain decrease in the anthropometric parameters body weight and waist circumference (associated with the modification of the unwanted habits).

The counseling intervention is the core of the multi-component remote care model, which also includes counseling through text messages, the purveyance of educational material, and self-monitoring equipment (pedometers and measuring tape for patients to check their waist circumference). The calls are made by professionals working at health centers who have been trained to apply theories on behavioral change and decision-making. Phone counseling are conducted at least once a month. Three different types of counseling are included: (a) Welcome: aimed at exploring the factors that promote behavioral change and the goals that the patient must reach to deal with prediabetes; (b) Follow-up: aimed at accompanying the patient and/or monitoring the attainment of goals associated with the desired behavioral change, (c) Completion: for closing the intervention process, reinforcing achievements, and inviting the patient to maintain the behavioral changes made. Short Message Service (SMS) counseling is aimed at providing information and encouraging the patient to change his/her behavior in terms of nutrition and physical activity. Messages are sent weekly and are related to the topics referred to in counseling sessions. The educational material and equipment --respectively-- seek to provide additional information and foster the habit of self-monitoring progress and/or reversions in the change process.

A randomized clinical study was designed, including a sample of 70 (both groups) people diagnosed with prediabetes and altered BMI, registered in 5 primary care centers in the La Florida commune, Santiago, Chile. The intervention will last 6 months. The control group will receive usual care from health centers consisting of an indication of physical activity and healthy eating recommendations, as well as referral to Dietitian if appropriate, an invitation to participate in educational activities at health centers and periodic inspection appointments. Apart from the usual care provided in health centers, the intervention group will also receive the four components of the remote care model. Pre and post intervention measurements will be applied. At the end of the intervention (after post-measurement) control group participants will be invited to participate in an educational workshop to improve eating practices and physical activity, and will receive educational materials generated by this project, thus ensuring the principle of equity in the project's development. For the intervention group, the program is expected to lead to increased knowledge on prediabetes, increment in physical activity, improvement of clinical and anthropometric parameters as well as of eating habits, all of these are non expected results for the control group.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes diagnosis
* 25- 34 Body Mass Index
* cellphone

Exclusion Criteria:

* Fasting blood glucose ≥ 126 (at the beginning of the intervention).
* Terminal chronic diseases
* Major cardiovascular problems (ie: angina pectoris, myocardial infarction, cerebrovascular accident)
* Severe psychiatric pathology
* Presence of another pathology which, for the doctor assessing the patient (at the beginning of the intervention), can be a contraindications to participate in the program.
* be pregnant
* To belong to private health system (called ISAPRE).

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Carola Pérez Ewert, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (5):
- Chile (5):
  - Centro de Salud Familiar Los Castaños, Santiago, Región Metropolitanta
  - Centro de Salud Santa Amalia, Santiago, Santiago Metropolitan
  - Centro de Salud Familiar Villa O'Higgins, Santiago, Santiago Metropolitan
  - Centro de Salud Familiar Fernando Maffioletti-Alvo, Santiago, Santiago Metropolitan
  - Centro de Salud Familiar Los Quillayes, Santiago, Santiago Metropolitan

RESULTS

PARTICIPANT FLOW:
Groups:
- Multicomponent Remote Care Model: Multicomponent remote care model: A remote intervention based on counseling (telephone-based) was implemented. This counseling intervention is the core of the multi-component model, which also includes counseling through text messages, the purveyance of educational material, and self-monitoring equipment (pedometer and measuring tape to check waist circumference). The phone counseling was made by professionals working at health centers who have been trained to apply theories on behavioral change and decision-making. A Mean of 5 phone counseling calls were done by participant. Messages were sent weekly and are related to the topics referred to in phone counseling sessions. The educational material and equipment -respectively- sought to provide additional information and foster the habit of self-monitoring progress and/or reversions in the change process.
Period: Overall Study
Arm/Group | Multicomponent Remote Care Model | Usual Care
Started | 36 | 34
Completed | 33 | 32
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multicomponent Remote Care Model | Usual Care | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.78 (8.46) | 54.88 (8.59) | 52.77 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 46
  Male | 10 | 14 | 24
Region of Enrollment [Number; unit: participants]
  Chile | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight Parameter
Description: Patient's weight wil be measured in kilograms using scales.
Time Frame: baseline and post intervention (6 -9 months after the first phone counseling session)
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Multicomponent Remote Care Model | Usual Care
Number analyzed (Participants) | 33 | 32
kilograms | -.58 (2.98) | -.18 (2.47)

2. Secondary Outcome: Change From Baseline in Self Report of Physical Activity
Description: The level of physical activity reported by participants is measured using the Rapid Assessment Physical Activity Scale (RAPA; Tolpolski et al., 2006), in its version adapted for Chile. This instrument is made up by 9 dichotomous questions, which point to a physical activity level corresponding to the following categories: sedentary, under-active, under-active regular-light activities, under-active regular, and active, depending on the frequency and intensity of the physical activity done. The instrument adaptation process of the instrument is conducted as part of the present study.
Time Frame: baseline and post intervention (6 -9 months after the first phone counseling session)
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: Fasting Glucose will be measured through a blood sample. The samples will be processed by the Municipal Laboratory (Laboratorio Comunal), following the standard procedures established by their protocols:
  Method:Colorimetric - Hexokinase / Glucose 6-phosphate-DH. UV. Equipment: Siemens Dimension RXL. Normal Range: 70-100 mg/dL.
Time Frame: baseline and post intervention (6 -9 months after the first phone counseling session)
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Triglycerides
Description: It will be measured through a blood sample. The samples will be processed by the Municipal Laboratory (Laboratorio Comunal), following the standard procedures established by their protocols:
  Method:Colorimetric - GPO/PAP blank glycerol. Equipment: Siemens Dimension RXL. Normal Range: ≤ 150 mg/dL.
Time Frame: baseline and post intervention (6 -9 months after the first phone counseling session)
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Total Cholesterol
Description: It will be measured through a blood sample. The samples will be processed by the Municipal Laboratory (Laboratorio Comunal), following the standard procedures established by their protocols:
  Method: Colorimetric - CHOD/PAP.Equipment: Siemens Dimension RXL. Normal Range: ≤ 200 mg/dL
Time Frame: baseline and post intervention (6 -9 months after the first phone counseling session)
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline in Self Report of Dietary Practices
Description: The dietary practices reported by the participants will be measured with an instrument designed with this purpose in mind as part of the present study. The instrument is constituted by 17 items aimed at measuring the frequency of healthy and unhealthy eating. It was constructed on the basis of items present in the Diabetes Self Care Activities Measure (Toobert, Hampson, & Glasgow, 2000) and of others created by the Stanford Patient Education Research Center. Some of these items were used to measure dietary practices in Chilean populations diagnosed with Diabetes Mellitus (Lange et al., 2010)
Time Frame: baseline and post intervention (6 -9 months after the first phone counseling session)
Reporting Status: Not Posted

7. Secondary Outcome: Change of Baseline in Knowledge About Prediabetes
Description: A self-report questionnaire was developed to measure patients' knowledge about prediabetes, the risk factors for its appearance, and its treatment (or management). Is is made up by 18 items in which the person must say whether the statement presented is true or false. In addition, the instrument measures the subjective perception of the risk of developing diabetes (one item).
Time Frame: baseline and post intervention (6 -9 months after the first phone counseling session)
Reporting Status: Not Posted

8. Secondary Outcome: Change of Baseline in Waist Circumference
Description: Participants' waist circumference will be measured in centimeters using a measuring tape. The circumference will be measured at the highest part of the iliac crest (The Canadian Physical Activity, Fitness and Lifestyle approach, 2010)
Time Frame: baseline and post intervention (6 -9 months after the first phone counseling session)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During the intervention time frame
Arm/Group | Multicomponent Remote Care Model | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 2/36 | 0/34
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Multicomponent Remote Care Model (N=36) | Usual Care (N=34)
falls (Musculoskeletal and connective tissue disorders) | 2 | 0 — falls during physical activity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No